CLINICAL TRIAL: NCT05682937
Title: High Frequency Oscillatory Ventilation Combined With Intermittent Sigh Breaths in Neonate: Effect on Carbon Dioxide Level
Brief Title: HFOV With Intermittent Sigh Breaths in Neonate: Carbon Dioxide Level
Acronym: SighCO2
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The duration of study was planned only 1 year owing to time constraints. Although the targeted sample size was not achieved, but the results showed significant difference between two interventions.
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Anucha Thatrimontrichai, Office of Human Research Ethics Unit, Prince of Songkla University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SighPSU
Record Dates: First submitted 2022-12-26; First posted 2023-01-12 (Actual); Results first posted 2025-01-29 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: High-Frequency Ventilation
Keywords: Carbon Dioxide; High-Frequency Ventilation; Sigh Breath; Newborn

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HFOV-sigh mode (Experimental): HFOV-sigh setting both brands of ventilator (SLE6000 and Drager Babylog VN500): setting (frequency [Hz], mean airway pressure [MAP], delta pressure [dP]) same as HFOV, set sigh RR 3 breath/min, Sigh inspiratory time [Ti] = 1 sec, Sigh peak inspiratory pressure [PIP] = (MAP+5, maximum 30) cm H2O, Slope sigh 0.5.
  Interventions: Device: HFOV-sigh

INTERVENTIONS:
Device: HFOV-sigh — HFOV-sigh setting both SLE6000 and Drager Babylog VN500: setting (Hz, MAP, delta pressure) same as HFOV, set sigh RR 3 breath/min, Sigh Ti = 1 sec, Sigh PIP = (MAP+5, maximum 30) cm H2O, Slope sigh 0.5.
  Other Names: HFOV-sigh application from both brands of ventilator (SLE6000 and Drager Babylog VN500)

SUMMARY:
The goal of this clinical trial is to the short-term effects of sigh breaths during High-frequency oscillatory ventilation (HFOV) in neonate undergoing mechanical ventilation. From meta-analysis, It revealed HFOV in neonates could reduce chronic lung disease or death rather than conventional ventilation.

The main question it aims to answer is: Do sigh breaths augment restoring lung volume and ventilation (CO2 level) in intubated neonate with HFOV? Participants will be applied sigh breaths (HFOV-sigh) during on HFOV. Researchers will compare HFOV-sigh mode to see if CO2 level (before-after intervention).

DETAILED DESCRIPTION:
Sample size calculation (before and after intervention: two dependent mean)

* alpha = 0.05, beta = 0.2,
* Delta = 1.9, SD. = 4.35
* Calculated sample size = 42
* increase sample size if loss follow up 20%
* Final sample size (n) = 50

Subgroup analysis for

* preterm neonates
* very preterm or very low birth weight neonates
* extremely preterm or extremely low birth weight neonates

ELIGIBILITY:
Inclusion Criteria:

* Preterm and term neonate (gestational age 24-41 weeks) with postnatal age less than 28 days
* Already ventilated with high frequency ventilation at least 1 hours
* An umbilical or peripheral arterial catheterization was available

Exclusion Criteria:

* Previous or current pulmonary air leaks (pulmonary interstitial emphysema, pneumothorax, pneumomediastinum, and pneumopericardium)
* Heterogeneous lung disease including MAS, congenital diaphragmatic hernia
* Suspected lung hypoplasia
* Suspected or confirmed intraventricular hemorrhage grade III-IV
* Suspected or confirmed hypoxic ischemic encephalopathy or 5-min Apgar score less than 3
* Hemodynamic instability despite using inotrope(s)
* Arterial pCO2 level less than 45 mm Hg or more than 70 mm Hg before intervention
* Need a new arterial puncture for samples both before and after interventions
* Moribund status
* Parents' decision not to participate

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2023-01-12 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anucha Thatrimontrichai, MD, Principal Investigator — Prince of Songkla University
Locations (1):
- Songklanagarind Hospital, Prince of Songkla University, Hat Yai, Changwat Songkhla, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cools F, Askie LM, Offringa M, Asselin JM, Calvert SA, Courtney SE, Dani C, Durand DJ, Gerstmann DR, Henderson-Smart DJ, Marlow N, Peacock JL, Pillow JJ, Soll RF, Thome UH, Truffert P, Schreiber MD, Van Reempts P, Vendettuoli V, Vento G; PreVILIG collaboration. Elective high-frequency oscillatory versus conventional ventilation in preterm infants: a systematic review and meta-analysis of individual patients' data. Lancet. 2010 Jun 12;375(9731):2082-91. doi: 10.1016/S0140-6736(10)60278-4. PMID 20552718
- [Result] Cools F, Offringa M, Askie LM. Elective high frequency oscillatory ventilation versus conventional ventilation for acute pulmonary dysfunction in preterm infants. Cochrane Database Syst Rev. 2015 Mar 19;2015(3):CD000104. doi: 10.1002/14651858.CD000104.pub4. PMID 25785789
- [Result] Courtney SE, Durand DJ, Asselin JM, Hudak ML, Aschner JL, Shoemaker CT; Neonatal Ventilation Study Group. High-frequency oscillatory ventilation versus conventional mechanical ventilation for very-low-birth-weight infants. N Engl J Med. 2002 Aug 29;347(9):643-52. doi: 10.1056/NEJMoa012750. PMID 12200551
- [Result] Hoch B, Bernhard M, Hinsch A. Different patterns of sighs in neonates and young infants. Biol Neonate. 1998;74(1):16-21. doi: 10.1159/000014006. PMID 9657665
- [Result] Jost K, Latzin P, Fouzas S, Proietti E, Delgado-Eckert EW, Frey U, Schulzke SM. Sigh-induced changes of breathing pattern in preterm infants. Physiol Rep. 2015 Nov;3(11):e12613. doi: 10.14814/phy2.12613. PMID 26564066
- [Result] Davis GM, Moscato J. Changes in lung mechanics following sighs in premature newborns without lung disease. Pediatr Pulmonol. 1994 Jan;17(1):26-30. doi: 10.1002/ppul.1950170106. PMID 8108173
- [Result] Qureshi M, Khalil M, Kwiatkowski K, Alvaro RE. Morphology of sighs and their role in the control of breathing in preterm infants, term infants and adults. Neonatology. 2009;96(1):43-9. doi: 10.1159/000201738. Epub 2009 Feb 10. PMID 19204409
- [Result] Patroniti N, Foti G, Cortinovis B, Maggioni E, Bigatello LM, Cereda M, Pesenti A. Sigh improves gas exchange and lung volume in patients with acute respiratory distress syndrome undergoing pressure support ventilation. Anesthesiology. 2002 Apr;96(4):788-94. doi: 10.1097/00000542-200204000-00004. PMID 11964584
- [Result] Mauri T, Eronia N, Abbruzzese C, Marcolin R, Coppadoro A, Spadaro S, Patroniti N, Bellani G, Pesenti A. Effects of Sigh on Regional Lung Strain and Ventilation Heterogeneity in Acute Respiratory Failure Patients Undergoing Assisted Mechanical Ventilation. Crit Care Med. 2015 Sep;43(9):1823-31. doi: 10.1097/CCM.0000000000001083. PMID 25985386
- [Result] Massaro GD, Massaro D. Morphologic evidence that large inflations of the lung stimulate secretion of surfactant. Am Rev Respir Dis. 1983 Feb;127(2):235-6. doi: 10.1164/arrd.1983.127.2.235. PMID 6687518
- [Result] Nacoti M, Spagnolli E, Bonanomi E, Barbanti C, Cereda M, Fumagalli R. Sigh improves gas exchange and respiratory mechanics in children undergoing pressure support after major surgery. Minerva Anestesiol. 2012 Aug;78(8):920-9. Epub 2012 Apr 27. PMID 22531559
- [Result] Bonacina D, Bronco A, Nacoti M, Ferrari F, Fazzi F, Bonanomi E, Bellani G. Pressure support ventilation, sigh adjunct to pressure support ventilation, and neurally adjusted ventilatory assist in infants after cardiac surgery: A physiologic crossover randomized study. Pediatr Pulmonol. 2019 Jul;54(7):1078-1086. doi: 10.1002/ppul.24335. Epub 2019 Apr 19. PMID 31004420
- [Result] Poets CF, Rau GA, Neuber K, Gappa M, Seidenberg J. Determinants of lung volume in spontaneously breathing preterm infants. Am J Respir Crit Care Med. 1997 Feb;155(2):649-53. doi: 10.1164/ajrccm.155.2.9032208.
- [Result] Sindelar R, Nakanishi H, Stanford AH, Colaizy TT, Klein JM. Respiratory management for extremely premature infants born at 22 to 23 weeks of gestation in proactive centers in Sweden, Japan, and USA. Semin Perinatol. 2022 Feb;46(1):151540. doi: 10.1016/j.semperi.2021.151540. Epub 2021 Nov 10. PMID 34872750

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Ninety-four infants were assessed for eligibility; 64 were excluded because of previous or current pulmonary air leaks (n = 3), heterogeneous lung diseases (n = 7), suspected or confirmed grade III-IV intraventricular hemorrhage (n = 1), hemodynamic instability despite using an inotrope (n = 15), PaCO2 level < 45 or > 70 mm Hg before intervention (n = 30), moribund status (n = 7), and parents' decision not to participate (n = 1). Thirty participants were finally enrolled.
Groups:
- HFOV-sigh Mode: HFOV-sigh setting both SLE6000 and Drager Babylog VN500: setting (Hz, MAP, delta pressure) same as HFOV, set sigh RR 3 breath/min, Sigh Ti = 1 sec, Sigh PIP = (MAP+5, maximum 30) cm H2O, Slope sigh 0.5.
Period: Overall Study
Arm/Group | HFOV-sigh Mode
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | HFOV-sigh Mode
Number analyzed (Participants) | 30
Age, Continuous [Median (Inter-Quartile Range); unit: day] | 1.88 [0.87 to 3.79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 30
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Gestational age [Mean (Standard Deviation); unit: weeks] | 33.6 (4.1)
Birth weight [Mean (Standard Deviation); unit: grams] | 2305 (853)

OUTCOME MEASURES:

1. Primary Outcome: Arterial pCO2 Level
Description: ABL800 BASIC (Radiometer Medical ApS™, Denmark) analyzed all blood gas samples within 1 min after collection. The blood gas machine was auto-calibrated every 4 h by trained specialists every day.
Time Frame: before sigh (baseline) and after sigh (2 hours)
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | HFOV-sigh Mode
Number analyzed (Participants) | 30
mm Hg
  HFOV before sigh | 48.8 (3.1)
  HFOV after sigh | 45.2 (6.6)

2. Secondary Outcome: Oxygenation
Description: oxygen index (oxygen index = mean airway pressure x FiO2 / PaO2), higher scores mean a worse outcome, no unit of scale.
Time Frame: before sigh (baseline) and after sigh (2 hours)
Population: oxygen index = mean airway pressure x FiO2 / PaO2
Measure: Median (Inter-Quartile Range); unit: no unit
Arm/Group | HFOV-sigh Mode
Number analyzed (Participants) | 30
no unit
  HFOV before sigh | 3.06 [2.48 to 4.26]
  HFOV after sigh | 2.95 [2.37 to 3.83]

3. Secondary Outcome: Mean Airway Pressure
Description: Mean Airway Pressure (MAP), cmH2O
Time Frame: 2 hours after sigh breaths
Population: the frequency of each MAP level was presented by the count of participants
Measure: Count of Participants; unit: Participants
Arm/Group | HFOV-sigh Mode
Number analyzed (Participants) | 30
Participants
  MAP = 7 cmH2O | 5
  MAP = 8 cmH2O | 12
  MAP = 9 cmH2O | 8
  MAP = 10 cmH2O | 4
  MAP = 13 cmH2O | 1

ADVERSE EVENTS:
Time Frame: 2 hours
Arm/Group | HFOV-sigh Mode
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-28): https://cdn.clinicaltrials.gov/large-docs/37/NCT05682937/Prot_SAP_000.pdf